CLINICAL TRIAL: NCT07210268
Title: Temporal Interference Methods for Addiction Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joshua Brown, PHD, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27333; 1R21DA062805-01 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Nicotine Use Disorder; Substance Use Disorders
Keywords: Nicotine Addiction; Non-invasive deep brain stimulation; Substance Use Disorders; Temporal Interference Stimulation; BOLD Activation
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: temporal interference stimulation to the nucleus accumbens, temporal interference stimulation to the anterior insula, or sham stimulation.
Who Masked: Participant
Masking Description: Participants will receive either active or sham stimulation with ramping protocols designed to mimic sensory experience across conditions. Participants are blinded to condition, and self-reported outcomes are collected through blinded survey methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- TI Stimulation - Nucleus Accumbens (Experimental): Participants in this arm will receive 60 minutes of temporal interference (TI) stimulation targeted to the nucleus accumbens (NAcc). TI will be delivered using two electrode sets, with placement determined to optimize stimulation of this region. Stimulation will use up to 2 mA per electrode at carrier frequencies of 2000 Hz and 2020 Hz, producing a 20 Hz beat frequency. Craving ratings will be collected every 10 minutes, and nicotine vapor use will be measured in real time.
  Interventions: Device: TI-NDBS
- TI Stimulation - Anterior Insula (Experimental): Participants in this arm will receive 60 minutes of temporal interference (TI) stimulation targeted to the anterior insula (AI). TI will be delivered using two electrode sets, with placement determined to optimize stimulation of this region. Stimulation will use up to 2 mA per electrode pair at carrier frequencies of 2000 Hz and 2020 Hz, producing a 20 Hz beat frequency. Craving ratings will be collected every 10 minutes, and nicotine vapor use will be measured in real time.
  Interventions: Device: TI-NDBS
- Sham Stimulation (Sham Comparator): Participants in this arm will receive sham temporal interference (TI) stimulation that mimics the initial sensation of active stimulation. The current will ramp up over 30 seconds and immediately ramp back down, with no sustained current. This procedure controls for sensory experience and participant expectations. Electrode placement will mirror that used in the active conditions. Participants will complete the same craving assessments and use the same custom vape device as in the experimental arms.
  Interventions: Device: Sham TI-NDBS

INTERVENTIONS:
Device: TI-NDBS — In the active TI-NDBS condition, participants receive transcranial stimulation for 60 minutes through scalp electrodes using temporal interference (TI). Two electrode sets deliver high-frequency alternating currents (e.g., 2000 Hz and 2020 Hz), generating a 20 Hz beat frequency at depth to stimulate targeted brain regions. Stimulation is delivered in six 10-minute blocks with 30-second ramp-up and ramp-down periods to minimize discomfort. Electrode configurations differ by group to target either the nucleus accumbens or anterior insula, based on finite element modeling. The maximum current is up to 2 mA per electrode, and no single region receives more than 2 mA.
  Other Names: Temporal Interference Non-invasive Deep Brain Stimulation
  Arms: TI Stimulation - Anterior Insula; TI Stimulation - Nucleus Accumbens
Device: Sham TI-NDBS — This is the control condition in which participants will receive sham stimulation for 60 minutes.
  Arms: Sham Stimulation

SUMMARY:
This clinical study is testing whether a new non-invasive brain stimulation method, called temporal interference (TI), can reduce nicotine cravings and usage in people who vape. TI delivers mild electrical currents to the scalp in a way that targets deep brain areas involved in addiction, without the need for surgery.

In this randomized controlled trial, participants will be assigned to one of three groups: TI stimulation to the nucleus accumbens, TI stimulation to the anterior insula, or a placebo (sham) condition. Each participant will attend a single stimulation session after 8 hours of nicotine abstinence and will use a custom vape device that measures real-time nicotine inhalation. Craving levels will be reported during and after the session.

The study aims to determine whether TI to the insula or nucleus accumbens is more effective at decreasing cravings and nicotine inhalation, and whether either is more effective than sham stimulation. For one week after the session, participants will use a smartphone app to track nicotine use and cravings. The primary hypothesis is that TI stimulation to deep brain regions will reduce both nicotine craving and actual use, immediately after stimulation and over the following week, compared to the sham condition.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) are difficult to treat effectively, with high relapse rates despite behavioral and pharmacological interventions. Previous clinical and case studies have shown that direct stimulation of deep brain regions-including the nucleus accumbens (NAcc) and anterior insula (AI)-can produce rapid, sustained reductions in addictive behaviors. Deep brain stimulation (DBS) of the NAcc has resulted in remission of opioid and alcohol use, while disruption of the AI has led to spontaneous loss of cigarette addiction. Although highly effective, DBS is invasive, expensive, and inaccessible to most patients. This randomized controlled clinical trial will evaluate whether temporal interference non-invasive deep brain stimulation (TI-NDBS) to the NAcc or AI can modulate deep brain activity and reduce nicotine craving and use in individuals who vape nicotine. TI uses two high-frequency electrical currents that intersect to create a low-frequency envelope capable of stimulating deep brain structures while sparing the overlying cortex. Pilot studies conducted by the investigators have shown that TI can safely and effectively activate the NAcc, as confirmed by increased BOLD signal during fMRI. In this study, 120 to 150 nicotine-dependent adults will be randomized to receive TI to the NAcc, TI to the AI, or sham stimulation. All participants will abstain from nicotine for at least 8 hours prior to the session, then undergo 60 minutes of stimulation while using a custom vape device that measures vapor inhalation in real time. Craving will be self-reported every 10 minutes. The primary outcome is a reduction in craving or nicotine use during the stimulation session. Secondary outcomes include changes in craving and use over the following week, assessed via ecological momentary assessment (EMA) three times daily using a smartphone app. Participants will also complete pre- and post-session assessments of cognitive function, emotional state, and stimulation experience. TI stimulation will be delivered with gradual current ramping to reduce discomfort, and previous pilot data support its tolerability. Findings from this study will provide early evidence of the safety and efficacy of TI-NDBS as a novel, low-cost, and scalable treatment for nicotine dependence, with potential applications in other addiction and psychiatric disorders involving deep brain circuitry.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 50
* Nicotine dependent and vape at least 15 mg nicotine per day
* Must have a phone with internet access
* Participants must have at least a 6th grade education and be able to speak and read English

Exclusion Criteria:

* History of seizures, seizure disorders, or familial history of seizure disorders
* History of intractable migraine or complicated migraine syndromes
* History of suicide attempts or active suicidal ideation (past month)
* History of cardiac arrhythmias, prolonged QT, pacemakers, or cardiovascular disorders
* Hypertension with systolic BP >150mmHgCentral nervous system structural lesions (tumors, MS, strokes, etc.)
* Active neuropsychiatric disorders (schizophrenia, bipolar, active psychosis, dementia, etc.)
* History of head trauma with loss of consciousness, skull fractures, subdural hematomas
* Active opioid, cocaine, and/or methamphetamine use
* Active severe cannabis use disorder
* Active alcohol use disorder or history of alcohol withdrawal
* Metal implants in the head or under the scalp (excluding dental implants)
* Current smoking cessation treatment or medications affecting reward processing
* Pregnancy

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in Nicotine Craving From Baseline to End of Stimulation Session | Baseline to 60 minutes post-stimulation initiation (during the single stimulation session)
  Nicotine craving will be assessed using a 1-10 Likert scale (1 = no craving, 10 = extremely strong craving) administered every 10 minutes during the 60-minute temporal interference (TI) stimulation session. The primary outcome is the change in self-reported craving from baseline (pre-stimulation) to the final rating at the 60-minute time point. This measure will assess the immediate effect of TI stimulation targeting either the nucleus accumbens or anterior insula on nicotine craving relative to sham stimulation.
Change in Nicotine Vapor Inhalation Volume From Baseline to End of 60-Minute Stimulation Session | Baseline to 60 minutes post-stimulation initiation
  Nicotine use will be assessed using a custom vape device that continuously measures the volume of inhaled vapor during the 60-minute stimulation session. The primary outcome is the change in total vapor volume compared to baseline, assessed across all three groups (NAcc, anterior insula, and sham).

SECONDARY OUTCOMES:
Change in Self-Reported Nicotine Craving Over 7-Day Post-Stimulation Period | Daily for 7 days post-stimulation
  Participants will report nicotine craving levels three times daily using ecological momentary assessment (EMA) via a smartphone app for seven days following the stimulation session. Ratings will use a 1-10 Likert scale, and group differences will be analyzed to assess lasting effects of stimulation.
Change in Self-Reported Nicotine Use Frequency Over 7-Day Post-Stimulation Period | Daily for 7 days post-stimulation
  Participants will self-report frequency of nicotine vaping or cigarette use three times daily via EMA for 7 days following the stimulation session. Daily use will be compared across groups to assess sustained effects on nicotine consumption.

OTHER OUTCOMES:
Change in Cognitive Function (Digit Span Test) From Pre- to Post-Stimulation | Immediately before to 10 minutes after stimulation session
  Cognitive function will be assessed before and after stimulation using the Digit Span subtest from the Wechsler Adult Intelligence Scale (WAIS-IV). This will evaluate short-term effects of TI stimulation on memory and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brown, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modak P, Fine J, Colon B, Need E, Cheng H, Hulvershorn L, Finn P, Brown JW. Temporal interference electrical neurostimulation at 20 Hz beat frequency leads to increased fMRI BOLD activation in orbitofrontal cortex in humans. Brain Stimul. 2024 Jul-Aug;17(4):867-875. doi: 10.1016/j.brs.2024.07.014. Epub 2024 Jul 24. PMID 39059712
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Publisher Correction: Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. No abstract available. PMID 37957321
- [Background] Naqvi NH, Rudrauf D, Damasio H, Bechara A. Damage to the insula disrupts addiction to cigarette smoking. Science. 2007 Jan 26;315(5811):531-4. doi: 10.1126/science.1135926. PMID 17255515
- [Background] Wessel MJ, Beanato E, Popa T, Windel F, Vassiliadis P, Menoud P, Beliaeva V, Violante IR, Abderrahmane H, Dzialecka P, Park CH, Maceira-Elvira P, Morishita T, Cassara AM, Steiner M, Grossman N, Neufeld E, Hummel FC. Noninvasive theta-burst stimulation of the human striatum enhances striatal activity and motor skill learning. Nat Neurosci. 2023 Nov;26(11):2005-2016. doi: 10.1038/s41593-023-01457-7. Epub 2023 Oct 19. PMID 37857774
- [Background] Joutsa J, Moussawi K, Siddiqi SH, Abdolahi A, Drew W, Cohen AL, Ross TJ, Deshpande HU, Wang HZ, Bruss J, Stein EA, Volkow ND, Grafman JH, van Wijngaarden E, Boes AD, Fox MD. Brain lesions disrupting addiction map to a common human brain circuit. Nat Med. 2022 Jun;28(6):1249-1255. doi: 10.1038/s41591-022-01834-y. Epub 2022 Jun 13. PMID 35697842
- See also: NIH Reporter Project Page — https://reporter.nih.gov/project-details/11116538